CLINICAL TRIAL: NCT06400862
Title: Treating Patients With Traumatic Chondral Lesions With Autologous Bone Marrow Cells Derived Engineered Tissues - Engineered Osteochondral Tissue
Acronym: TCL-aMSC-eOCT
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Chan Pui Barbara, Professor, Chinese University of Hong Kong
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: eOCT
Record Dates: First submitted 2024-03-09; First posted 2024-05-06 (Actual); Last update posted 2024-05-06 (Actual); Status verified 2024-05

CONDITIONS: Traumatic Cartilage Injury
Keywords: traumatic knee cartilage injury

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- eOCT Treatment (Experimental): In a pre-treatment visit, bone marrow aspiration will be conducted to harvest autologous bone marrow for mesenchymal stem/stromal cells (MSCs) isolation for subsequent eOCT manufacturing. Cartilage lesion will be addressed in the treatment visit by delivering eOCT through arthroscopic surgery roughly 13 weeks after the pre-treatment visit.
  Interventions: Combination Product: eOCT implantation

INTERVENTIONS:
Combination Product: eOCT implantation — eOCT is regarded as an Advanced Therapy Product (ATP).

SUMMARY:
The objective of the study is to establish the safety profile of the autologous engineered osteochondral tissues (eOCT) in treating traumatic chondral lesions in patients.

DETAILED DESCRIPTION:
TCL-aMSC- eOCT is a single arm first-in-human trial designed to establish the safety profile of autologous tissue engineered osteochondral tissue (eOCT) in patients with traumatic chondral lesions. Patient selection will base on medical records, especially MRI results, and other criteria. Patient enrollment and informed consent will be conducted at the baseline visit. In a pre-treatment visit, bone marrow aspiration will be conducted to harvest autologous bone marrow for mesenchymal stem/stromal cells (MSCs) isolation and subsequent eOCT manufacturing. Cartilage lesion will be repaired in the treatment visit by delivering eOCT through arthroscopic surgery roughly 13 weeks after the pre-treatment visit. Rehabilitation will be conducted post-implantation. Multiple follow-up visits will be conducted up to 24 months post-implantation, data including adverse events, clinical and functional scoring and blood tests will be collected during each follow-up visit. Radiological assessment such as magnetic resonance imaging (MRI) will be conducted regularly until the end of the study.

ELIGIBILITY:
Inclusion Criteria:

* Age: Subjects who are in the age range of 18-60 years
* Location: Single symptomatic cartilage defect on medial or lateral femoral condyle
* Size & Containment: Contained single focal cartilage lesion of size ~1-4 cm square
* Grading: Cartilage damage ICRS/Outerbridge grade III/IV reaching subchondral bone (As diagnosed by MRI)
* Conservative treatments failed (for > 4 months)

Exclusion Criteria:

Disease Factor---

* Previous cartilage repair surgery (OATS or ACI/MACI) in the index knee
* Previous injectional treatments such as HA/PRP/stem cell in the index knee within 3 months before informed consent
* Presence of a clinically relevant patellofemoral cartilage lesion in the index knee (patella/trochlea/both)
* Inflammatory joint disease (specific or non-specific arthritis)
* Metabolic diseases (gout or rheumatism)
* Advanced Osteoarthritis (Radiologically apparent degenerative joint disease in the target knee as determined by Kellgren & Lawrence Grade >2)
* Osteochondritis dissecans
* Multiple or uncontained lesions as detected by MRI or arthroscopy
* Uncorrected ligament deficiency
* Uncorrected varus or valgus malalignment exceeding 5°
* Ongoing Infection or skin diseases at target knee joint
* Significant meniscal loss

Patient Factor---

* Subjects who are not able or not willing to give voluntary, written informed consent to participate in this study
* Skeletal immaturity
* Female subjects who are pregnant or lactating
* Body mass index > 30 kg/m2
* Malignancy
* Steroid therapy by systemic or intra-articular route within the last 60 days before informed consent or intramuscular or oral steroids within the last 30 days before informed consent
* Contraindications to MR imaging
* Drug addiction (including narcotic, anesthetic or alcohol addiction)
* Patients who are at higher risk for post-surgical bleeding (e.g., bleeding disorder; taking anticoagulants except low dose aspirin
* Patients who are at higher risk for post-surgical infection (e.g., taking immunosuppressants; have a severe infection or a history of serious infection)
* Known allergy to porcine/bovine collagen
* Any concomitant painful or disabling disease of the spine, hips, or lower limbs that would interfere with evaluation of the afflicted knee
* Patients with human immunodeficiency virus, hepatitis, or syphilis
* Any clinically significant or symptomatic vascular or neurologic disorder of the lower extremities
* Poor general health condition as judged by investigator
* Unable to do follow up

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 9 (Estimated)
Dates: Start 2024-02-26 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Safety Outcomes | From subject enrollment to 24 months after the eOCT implantation.
  Incidence of Adverse events/ Serious adverse events (AEs/SAEs).
  To establish the safety profile of the autologous engineered osteochondral tissues (eOCT) from the data collected on adverse events/ serious adverse events.

SECONDARY OUTCOMES:
Visual Analogue Scale (VAS) | From subject enrollment to 24 months after the eOCT implantation.
  The Visual Analogue Scale (VAS) measures pain intensity of the participants, where 0 represents no pain and 10 represents the worst pain imaginable.
Knee Injury and Osteoarthritis Outcome Score (KOOS) | From subject enrollment to 24 months after the eOCT implantation.
  KOOS is a specialized tool designed to gather patients' perspectives on their knee and associated problems. It evaluates both short-term and long-term consequences of knee injury and has five subscales to assess the knee: pain symptoms, activities of daily living, sport and recreation function and knee-related quality of life.
The Western Ontario and McMaster University Osteoarthritis index (WOMAC) | From subject enrollment to 24 months after the eOCT implantation.
  WOMAC is a widely used questionnaires to evaluate the functional condition of participant's hip and knee osteoarthritis. It includes 3 subscales: pain, stiffness, and physical functioning of the joints, and assess the activities of daily living, functional mobility, gait, general health and the quality of life.
World Health Organization Quality of Life Instruments (WHOQOL-BREF) | From subject enrollment to 24 months after the eOCT implantation.
  WHOQOL-BREF is a quality-of-life scale developed through the World Health Organization which contains 26 items.
Short-Form- 36 (SF-36) | From subject enrollment to 24 months after the eOCT implantation.
  The SF-36 health survey has 36 questions to measure the functional health and general well-being of a participant. It is a reliable and validated measure that summarizes the participants' physical and mental health.
Kellgren and Lawrence (K&L) grading | From subject enrollment to 24 months after the eOCT implantation.
  K&L grading is a common method of classifying the severity of osteoarthritis (OA) using five grades.
Magnetic Resonance Observation of Cartilage Repair Tissue (MOCART) Score 2.0 | From subject enrollment to 24 months after the eOCT implantation.
  MOCART 2.0 scoring will occur by independent assessment to evaluate the cartilage repair tissue. The score is a 7-part and 24-item scoring system, also resulting in a final cartilage repair tissue score between 0 and 100 points; 0 points represent the worst imaginable score, 100 points represent the best imaginable score.
T2 mapping signal | From subject enrollment to 24 months after the eOCT implantation.
  The value T2 mapping signal represents continuous data of the T2 mapping signal intensity at the defect site relative to that of the surrounding uninjured cartilage, with arbitrary units, measuring the quality of the cartilage at the defect site.
Cartilage thickness | From subject enrollment to 24 months after the eOCT implantation.
  Cartilage thickness (mm) of cartilage lesion and neighboring normal cartilage measured by specific sequence.

CONTACTS AND LOCATIONS:
Overall Officials: Barbara Pui CHAN, PhD, Principal Investigator — Chinese University of Hong Kong
Locations (2):
- Hong Kong (2):
  - Queen Elizabeth Hospital, Jordon
  - Prince of Wales Hospital, Shatin

IPD SHARING:
Plan to Share IPD: No